CLINICAL TRIAL: NCT01757899
Title: Phase II, Randomized, Placebo-Controlled, Double-Blind Clinical Trial to Evaluate the Effects and Safety of Infusion of Low-Doses of Methylprednisolone in Early ALI and ARDS in Children
Brief Title: Effects and Safety of Infusion of Low-Doses of Methylprednisolone in Early ALI and ARDS in Children
Acronym: PEDALI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Technical problems
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Instituto de Puericultura e Pediatria Martagão Gesteira - IPPMG/UFRJ (Unknown); Instituto D'Or de Pesquisa (Unknown); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Fernanda Lima, MD Msc, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONEP 16487
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: ALI; Acute Lung Injury; ARDS; Acute Respiratory Distress Syndrome; Pediatric Critical Care Medicine; Inflammatory Response
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone Arm (Active Comparator): The patients in this arm will receive methylprednisolone, which is available in vials containing 125 mg/2mL after dilution, as it follows:
  Day 0 Loading dose 1 mg/kg IV bolus mixed in 5 mL NS (30 min) followed by continuous infusion Days 0 to 07 - 1 mg/kg/day mixed in 24cc NS and infused at 1 cc/hr Days 08 to 10 - 0.5 mg/kg/day mixed in 24cc NS and infused at 1 cc/hr Days 11 to 12 - 0.25 mg/kg/day Days 13 to 14 - 0.125 mg/kg/day
  Interventions: Drug: Methylprednisolone Arm
- Sterile Saline Arm (Placebo Comparator): Patients randomized to the control arm will receive sterile normal saline in an amount that would equal the total diluted dose of study drug (ie. if initial loading dose equals a total of 24 cc [methylprednisolone + diluting fluid], then the patient will receive 24 cc of sterile normal saline). Tapering doses will be equivalent to that of the study arm, so that investigators will remain blinded to therapy. The unblinded party will be composed of the research ARDS pharmacist. Five days after the patient is able to ingest medications, placebo is administered per os (PO) in one single daily equivalent dose. The placebo will be manipulated by the pharmacist as to resemble identical to the active drug.
  Interventions: Drug: Sterile Saline Arm

INTERVENTIONS:
Drug: Methylprednisolone Arm — Day 0 - Loading dose 1 mg/kg IV bolus mixed in 5 mL NS (30 min) followed by continuous infusion Days 0 to 07 - 1 mg/kg/day mixed in 24cc NS and infused at 1 cc/hr Days 08 to 10 - 0.5 mg/kg/day mixed in 24cc NS and infused at 1 cc/hr Days 11 to 12 - 0.25 mg/kg/day Days 13 to 14 - 0.125 mg/kg/day
  Other Names: Solumedrol
  Arms: Methylprednisolone Arm
Drug: Sterile Saline Arm — Patients randomized to the control arm will receive sterile normal saline in an amount that would equal the total diluted dose of study drug (ie. if initial loading dose equals a total of 24 cc [methylprednisolone + diluting fluid], then the patient will receive 24 cc of sterile normal saline). Tapering doses will be equivalent to that of the study arm, so that investigators will remain blinded to therapy. The unblinded party will be composed of the research ARDS pharmacist. Five days after the patient is able to ingest medications, placebo is administered per os (PO) in one single daily equivalent dose. The placebo will be manipulated by the pharmacist as to resemble identical to the active drug.
  Other Names: Saline
  Arms: Sterile Saline Arm

SUMMARY:
The purpose of this study is to investigate the effects of prolonged low-dose methylprednisolone infusion on pulmonary function (LIS and ventilation-free days), extra pulmonary organ function (PMODS score), inflammatory markers - RCP (Reactive C Protein), IL6 (Interleukine 6), TNFα (Tumor Necrosis Factor), IL8 (Interleukine 8), IL10 (Interleukine 10) and length of Pediatric Intensive Care Unit (PICU) stay in early ALI/ARDS in children.

DETAILED DESCRIPTION:
Scientific background. Dysregulated systemic inflammation - characterized by protracted elevation of inflammatory cytokines in the circulation - is a key pathogenetic mechanism for morbidity and mortality in ALI/ARDS, and is associated with tissue insensitivity and/or resistance to inappropriately elevated endogenous glucocorticoids. In one study, prolonged methylprednisolone treatment of ARDS patients resulted in rapid and sustained reduction in circulating and pulmonary levels of pro-inflammatory cytokines, chemokines, and procollagen.

Preliminary work. Two recent metanalysis evaluating the use of low doses of corticosteroids in acute lung injury/ARDS in adults reported a significant physiological improvement, a sizable reduction in duration of mechanical ventilation and ICU length of stay and reduction in mortality.

Hypothesis. We hypothesized that prolonged administration of low doses of methylprednisolone in pediatric ALI/ARDS is safe and downregulates systemic inflammation and leads to earlier resolution of pulmonary and extra pulmonary organ dysfunction and a reduction in duration of mechanical ventilation and ICU stay.

Objective. To investigate the effects of prolonged low-dose methylprednisolone infusion on pulmonary function (LIS and ventilation-free days), extra pulmonary organ function (PMODS score), inflammatory markers - RCP (Reactive C Protein), IL6 (Interleukine 6), TNFα (Tumor Necrosis Factor), IL8 (Interleukine 8), IL10 (Interleukine 10) and length of Pediatric Intensive Care Unit (PICU) stay in early ALI/ARDS in children.

Study design. Prospective randomized, placebo-controlled, double-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALI/ARDS within the first 72 hours based on all of the following criteria:

  * Respiratory failure requiring mechanical ventilation - via endotracheal intubation or noninvasive positive pressure ventilation;
  * Acute onset of bilateral pulmonary densities on chest radiograph in the context of appropriate predisposing injury or illness with no evidence of left ventricular failure;
  * Ratio of partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2:FiO2 ) ≤ 300 (criteria for ALI) or 200 (criteria for ARDS) with FiO2 ≥ 0,5 and PEEP = 5 cmH2O.
* To sign the Informed Consent to participate.

Exclusion Criteria:

* ALI/ARDS with more than 72 hours of diagnosis
* Failure to obtain written informed consent to participate in the study;
* Condition requiring > 0.5mg/Kg/day of prednisone equivalent (i.e., acute asthma or bronchopulmonary dysplasia)
* Patients enrolled in another experimental (interventional) protocol within the past 30 days, which might adversely impact on the results of this study as determined by the investigators;
* Primary or secondary neuromuscular dysfunction
* Patients using aminoglycosides combined with neuromuscular blockers
* Cardiopulmonary arrest within 7 days or anytime during present hospitalization prior to enrollment;
* Irreversible cessation of all brain function;
* Immunosuppression, including HIV+ status, history of bone marrow or solid organ transplantation, current malignancy, neutropenia, receiving cytotoxic therapy for any reason, and acute burn injury;
* Severe chronic liver disease (Child-Pugh Class C score > 10 points).

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Effects on pulmonary organ function | 24 months
  * a ≥ 1-point reduction in LIS by study day 7 or successful extubation by day 7
  * For patients remaining intubated on study day 7, improvement in lung function is defined as a 7-day LIS ≤ 2 (if initial LIS ≤ 2,9) or a 7-day LIS ≥ 2,5 (if initial LIS ≥ 3)
  Duration of mechanical ventilation defined as:
  * ventilator free days at 28 days of entry study
  * days of mechanical ventilation on day 28

SECONDARY OUTCOMES:
Effects on extra-pulmonary organ function | 24 months
  pediatric multiple organ dysfunction score (P-MODS) by study day 7
Effects on inflammatory process | 24 months
  Levels of CRP, TNFα, IL-6, IL-8, IL-10 by study day 7
Effects on hospitalization-related outcomes | 24 months
  Length of PICU stay

OTHER OUTCOMES:
Complications | 12 months
  Rate of new infections after study entry, defined as:
  * number of patients with new nosocomial infections
  * number of new nosocomial infections after study entry
Complications | 12 months
  Rate of potential complications associated with treatment, defined as:
  * number of patients developing hyperglycemia requiring insulin
  * pancreatitis (defined by elevated serum lipase level)
  * gastrointestinal bleeding
  * hypernatremia
  * behavioral disorders (clinical judgment and parents report)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Clara M Barbosa, Study Chair — Instituto D'Or de Pesquisa; Arnaldo P Barbosa, Study Director — Rio de Janeiro Federal University; Antonio José LA Cunha, Study Director — Rio de Janeiro Federal University; Fernanda Lima, Principal Investigator — Instituto D'Or de Pesquisa
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Sweeney RM, McAuley DF. Prolonged glucocorticoid treatment in acute respiratory distress syndrome - Authors' reply. Lancet. 2017 Apr 15;389(10078):1516-1517. doi: 10.1016/S0140-6736(17)30953-4. No abstract available. PMID 28422025